CLINICAL TRIAL: NCT03242980
Title: Short Adherence Intervention for Viral Re-suppression (SAVIR) Study: A Stepped Wedge Randomized Controlled Study to Assess the Effect of Standardized Adherence Counselling in Individuals With Unsuppressed Viral Load in Lesotho
Brief Title: Short Adherence Intervention for Viral Re-suppression
Acronym: SAVIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: SolidarMed (Other); Ministry of Health, Lesotho (Other Government); University of Basel (Other)
Responsible Party: Principal Investigator, Tracy Glass, Project Leader, Swiss Tropical & Public Health Institute
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: SAVIR
Record Dates: First submitted 2017-08-02; First posted 2017-08-08 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Adherence, Medication; HIV/AIDS
Keywords: HIV; Adherence; Viral re-suppression; Step-wedgged randomized trial
MeSH Terms: conditions — Medication Adherence; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: To ensure that the effect of this intervention is measured and to avoid a long delay in adopting the intervention, a stepped wedge design was chosen. In addition the study would thus not disrupt the on-going staggered roll-out of routine viral load provision to patients on ART at the 12 health facilities. Stepped wedge designs are a form of clustered study in which the intervention is delivered to groups rather than individuals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced adherence counseling (No Intervention): Individuals with elevated VL are required to attend a minimum of 2 session of enhanced adherence counselling performed at monthly intervals. A follow-up VL is done at 8 to 12 weeks after the first counselling session.
- Structured EAC plus SMS (Experimental): The behavioral intervention will consist of structured adherence counseling and a short text message (SMS). A culturally adapted graphical brochure was specifically developed to guide adherence-counselling for individuals with unsuppressed VL.
  Interventions: Behavioral: Structured adherence counseling

INTERVENTIONS:
Behavioral: Structured adherence counseling — Patients will undergo one standardized enhanced adherence counselling session. Counselling guidelines and a brochure were specifically developed to guide the adherence counselling for individuals with unsuppressed VL. All nurses at the health centres will be trained on the counselling prior to the cross-over to the intervention. The brochure was developed by culturally adapted by social scientists and contains only 3 key messages. The brochure will be given to the patient to take home.
  Four weeks after the adherence counselling session, a SMS will be sent to the patient reminding them to take their ART. The content of the text message will be anonymous to protect disclosure and discussed/agreed upon with the patient during the adherence counselling.
  Arms: Structured EAC plus SMS

SUMMARY:
In the era of test-and-treat, with anticipated high numbers of patients who will have unsuppressed viral load (VL) due to poor adherence, simple, short and standardized adherence interventions with documented efficacy will be needed. Achieving re-suppression in patients with unsuppressed VL is beneficial for the health of the individual, important to reduce the risk of transmission and has a direct cost implication because patients with sustained unsuppressed VL will ultimately be switched to more expensive 2nd-line regimens.

Information is still largely lacking on how to best address adherence problems among patients with unsuppressed VL. VL monitoring is recognized as a useful tool to reinforce adherence in patients with unsuppressed VL. The Lesotho Guidelines recommend redoing a VL 8-12 weeks after the first enhanced adherence counselling. To date no study has been published clearly demonstrating higher re-suppression rates after enhanced adherence counselling for patients with unsuppressed VL.

This project aims to test an adherence intervention for HIV-positive individuals on first-line ART who have an unsuppressed viral load. A step wedged study will be used to compare the effectiveness of a short, standardized adherence counselling followed by an SMS reminder to the standard of care (≥ 2 unstructured adherence counselling sessions) in terms of viral re-suppression rates and switches to 2nd line ART.

DETAILED DESCRIPTION:
Due to a lack of routine viral load (VL) monitoring in Lesotho until now, most health care workers in the districts lack the necessary information on how to manage patients with elevated viral loads. The CART-1 study found re-suppression rates of only 30% with only 70% returning for a second VL. From these estimates, it is clear that the current practice for managing these patients must be improved. A simple intervention has been designed that could be feasibly adapted at all health centres in Lesotho.

To ensure that the effect of this intervention is measured and to avoid a long delay in adopting the intervention, a stepped wedge design was chosen. In addition the study would thus not disrupt the on-going staggered roll-out of routine viral load provision to patients on ART at the 12 health facilities. Stepped wedge designs are a form of clustered study in which the intervention is delivered to groups rather than individuals. In this case, the cluster is the hospital or health centre. Each health centre will undergo a time period with the standard of care and then will be randomly selected to cross-over to the intervention at different time points, until all of the health centres have crossed-over to receive the intervention. Data on the endpoint will be collected continuously at all health centres. The use of a step wedged study is pragmatic - the intervention is offered to exert its expected benefits and research insight is a secondary aim. This innovative design will lead to much stronger evidence than observational studies.

Routine VL (viral load) monitoring started in Butha-Buthe hospital in December 2015, in Seboche Hospital in May 2016 and the remaining 10 health centres in June 2016. Once each hospital/health center has implemented routine VL monitoring for a least 12 weeks, the standardized adherence intervention will be rolled out to the hospitals/health centers in a randomized fashion. Every 12 weeks starting in May 2017, two hospitals/health centers will be randomly selected to start with the adherence intervention.

Randomization times will be separated by 12 weeks to allow for implementation and assessment of the intervention within each time period. Final data collection will occur in October 2018. All nurses at the centres will be trained in the standardized adherence counselling by an experienced professional counselor and an experienced ART nurse prior to the introduction of the intervention.

The tracing of patients who do not show up for adherence counselling sessions or confirmatory VL will be done according to the current system in use at the health centre (usually contact individual via village health worker or phone if available) and will remain the same during both the control and intervention period.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving VL monitoring at one of the 2 hospitals and 10 health centres in Butha-Buthe district
* Patients on first-line ART
* Patients with a VL≥ 1000 copies/mL after a minimum of 6 months on first-line ART

Exclusion Criteria:

* Patients receiving VL monitoring at a non-participating center in Butha-Buthe

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 928 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Re-suppression rates after one elevated viral load | Up to 16 weeks
  HIV viral load <1000 copies/ml

SECONDARY OUTCOMES:
Rates of switch to second-line ART | Up to 6 months
  Any switch to protease-inhibitor based ART
Major drug resistance mutations | 3 months after 1st elevated VL
  Presence of any major drug resistance mutation in those with 2nd elevated VL
Rates of attrition from care | 6 months
  No attendance at the clinic within 6 months after informing the patient about his/her first elevated VL
Rates of viral re-suppression | 6 months after switch
  In those who switched to 2nd line

CONTACTS AND LOCATIONS:
Overall Officials: Tracy R Glass, PhD, Principal Investigator — Swiss TPH; Niklaus Labhardt, MD, Study Chair — Swiss TPH
Locations (12):
- Lesotho (12):
  - Boiketsiso Health Center, Butha-Buthe
  - Linakeng Health Center, Butha-Buthe
  - Makhunoane Health Center, Butha-Buthe
  - Motete Health Center, Butha-Buthe
  - Muela Health Center, Butha-Buthe
  - Ngoajane Health Center, Butha-Buthe
  - Paballong, Butha-Buthe
  - Rampai Health Center, Butha-Buthe
  - Seboche, Butha-Buthe
  - St Paul Health Center, Butha-Buthe
  - St Peters Health Center, Butha-Buthe
  - Tsime Health Center, Butha-Buthe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Government of Lesotho: NATIONAL GUIDELINES ON THE USE OF ANTIRETROVIRAL THERAPY FOR HIV PREVENTION AND TREATMENT. Fifth Edition 2016.
- [Background] Conway B. The role of adherence to antiretroviral therapy in the management of HIV infection. J Acquir Immune Defic Syndr. 2007 Jun 1;45 Suppl 1:S14-8. doi: 10.1097/QAI.0b013e3180600766. PMID 17525686
- [Background] Bonner K, Mezochow A, Roberts T, Ford N, Cohn J. Viral load monitoring as a tool to reinforce adherence: a systematic review. J Acquir Immune Defic Syndr. 2013 Sep 1;64(1):74-8. doi: 10.1097/QAI.0b013e31829f05ac. PMID 23774877
- [Background] Jobanputra K, Parker LA, Azih C, Okello V, Maphalala G, Kershberger B, Khogali M, Lujan J, Antierens A, Teck R, Ellman T, Kosgei R, Reid T. Factors associated with virological failure and suppression after enhanced adherence counselling, in children, adolescents and adults on antiretroviral therapy for HIV in Swaziland. PLoS One. 2015 Feb 19;10(2):e0116144. doi: 10.1371/journal.pone.0116144. eCollection 2015. PMID 25695494
- [Background] Ministry of Health and Social Welfare Lesotho: National Guidelines For HIV Testing And Counselling. National Guidelines For HIV Testing And Counselling 2009.